CLINICAL TRIAL: NCT01797874
Title: Phase II Study of Pazopanib Maintenance for SCLC
Brief Title: Pazopanib Maintenance for SCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Myung-Ju Ahn, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-09-060-002
Record Dates: First submitted 2013-02-21; First posted 2013-02-25 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: SCLC
Keywords: pazopanib maintenance; efficacy; SCLC
MeSH Terms: interventions — pazopanib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pazopanib (Experimental): pazopanib maintenance after 4 cycles of etoposide/platinum in SCLC
  Interventions: Drug: Pazopanib
- placebo (Placebo Comparator): placebo after 4 cycles of etoposide/platinum chemotherapy in SCLC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pazopanib — Experimental
  Other Names: Votrient
  Arms: Pazopanib
Drug: Placebo — placebo arm
  Arms: placebo

SUMMARY:
To evaluate the efficacy of pazopanib maintenance after 1st line CTx for SCLC.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed SCLC
* no disease progression after 4 cycles of etoposide/platinum 1st-line therapy
* history of 4 cycles of etoposide/platinum 1st-line therapy
* between 21 days and 42 days since C4D1 of etoposide/platinum
* no symptomatic brain meta

Exclusion Criteria:

* poor hepatic, renal function

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea